CLINICAL TRIAL: NCT03884894
Title: PCR Technique of a Commercial Test and Blood Culture to Early Detect Sepsis in NICU
Brief Title: Neonatal Sepsis Diagnosis: ; PCR Commercial Technique and Blood Culture
Status: Completed | Type: Observational
Sponsor: Francesca Garofoli (Other)
Responsible Party: Sponsor-Investigator, Francesca Garofoli, Doctor, Fondazione IRCCS Policlinico San Matteo di Pavia
Organization: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Other Study IDs: IRCCSPSM/Eusepscreen/2015
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Sepsis
Keywords: neonatal sepsis; Blood culture; molecular assay
MeSH Terms: conditions — Sepsis; Neonatal Sepsis | interventions — Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- sepsis diagnosis by blood colture/molecular biology: fullterm/ preterm neonates hospitalized in NICU with suspect of sepsis
  Interventions: Diagnostic Test: molecular assay; Diagnostic Test: Blood culture

INTERVENTIONS:
Diagnostic Test: molecular assay — performed with blood culture simultaneously
  Other Names: "EuSepScreen lattanti" diagnostic kit
Diagnostic Test: Blood culture — performed with molecular assay simultaneously

SUMMARY:
Although advances in neonatal care have improved survival and reduced complications in preterm infants, sepsis still contributes significantly to mortality and in Neonatal Intensive Care Units (NICUs), in particular for very-low-birth-weight (VLBW, <1500 g) and extremely-low-birth-weight (ELBW, <1000g). Based on the timing of the infection neonatal sepsis has been classified into early-onset sepsis (EOS) and late-onset sepsis (LOS), with differences in the mode of transmission and predominant organisms. EOS is defined as onset in the first 3 days of life generally due to vertical transmission of bacteria from mothers to infants during the intrapartum period. LOS occurs after 3 days of life and it is attributed to pathogens acquired postnatally (horizontal transmission). Considering generally neonatal sepsis in Europe, 90% of the responsible bacteria resulted to be: Streptococcus agalactiae, Escherichia coli, Klebsiella pneumoniae, e Listeria monocytogenes. The diagnosis is difficult because clinical signs, particularly early in the course of disease, are subtle and nonspecific, and laboratory tests and blood culture are not always reliable. Moreover. blood culture (considered the 'gold standard) takes 48-72 hours for result. In fact the cultural method requires the presence of living and vital germs, depends on the volume of the sample - serious problem in neonatal population -, several hours are needed to process the sample, possibly resulting falsely negative in subjects undergoing concomitant antibiotic treatment or a false positive result can be found by contamination. The method based on molecular biology does not require living germs and, therefore, is not characterised by the sensitivity limitations. Such method can result to be extremely effective in patients receiving antibiotic therapy.

In the present study, when an infant has to undergone blood sample for bacteria culture to verify a possible sepsis, a residual blood (200µl) is processed in the same time using a kit based on molecular biology.

This kit is designed to obtain the highest sensitivity and specificity in the determination of most invasive bacterial diseases (meningitis, sepsis, pneumonia, etc.) affecting full-term, preterm infants to determine any presence of bacterial DNA belonging to all serotypes of Klebsiella pneumoniae, Escherichia coli, Streptococcus agalactiae and Listeria monocytogenes.

The target bacteria have been chosen on the basis of the current Italian epidemiological context, so as to include germs causing about 90% of the meningitis/sepsis cases among the neonatal population. The detection system can unmistakably identify the germ against which it is directed and without causing any cross-reaction with other germs or human DNA..

The results obtained with this method have demonstrated a 100% specificity (no false positive result) The sensitivity of this method compared with the cultural method has turned out to be twice as high.

The aim of the present study is to compare the efficacy of the blood culture method and the kit for molecular detection of bacterial DNA (all serotypes of Klebsiella pneumoniae, Escherichia coli, Streptococcus agalactiae and Listeria monocytogenes) considering the relevant epidemiology of our NICU, in order to verify the relative frequency of sepsis (EOS and LOS) caused by the target bacteria on the whole frequency of the bacteria responsible of all the sepsis in our ward.

DETAILED DESCRIPTION:
Neonatal sepsis remains one of the leading causes of morbidity and mortality both among term and preterm infants. Although advances in neonatal care have improved survival and reduced complications in preterm infants, sepsis still contributes significantly to mortality and in Neonatal Intensive Care Units (NICUs).in particular for very-low-birth-weight (VLBW, <1500 g) and extremely-low-birth-weight (ELBW, <1000g).The signs and symptoms of neonatal sepsis are non specific. These include fever or hypothermia, respiratory distress including cyanosis and apnea, feeding difficulties, lethargy or irritability, hypotonia, seizures, bulging fontanel... Based on the timing of the infection neonatal sepsis has been classified into early-onset sepsis (EOS) and late-onset sepsis (LOS), with differences in the mode of transmission and predominant organisms. EOS is defined as onset in the first 3 days of life generally due to vertical transmission of bacteria from mothers to infants during the intrapartum period. LOS occurs after 3 days of life and it is attributed to pathogens acquired postnatally (horizontal transmission). The epidemiology of neonatal sepsis is a changing landscape, nevertheless an increasing rates of EOS Escherichia coli sepsis, particularly among preterm infants, and Streptococcus group B (GBS), in particular S. agalactiae, - resulted to be 70% of the responsible microorganisms, In a study on 6215 infants admitted to National Institute of Child Health and Human Development (NICHD) Neonatal Research Network (NRN) centres, 70% of first episode late-onset infections were caused by gram-positive organisms, with coagulase-negative staphylococci accounting for 48% of the infections. Considering generally neonatal sepsis in Europe, 90% of the responsible bacteria resulted to be: Streptococcus agalactiae, Escherichia coli, Klebsiella pneumoniae, e Listeria monocytogenes. The diagnosis of neonatal sepsis is difficult because clinical signs, particularly early in the course of disease, are subtle and nonspecific, and laboratory tests and blood culture are not always reliable, moreover blood culture, (the 'gold standard) takes 48-72 hours or more for result. In fact the cultural method shows a number of weak points: it requires the presence of living and vital germs, it depends on the volume of the collected sample - serious problem in neonatal population -, several hours are needed to process the sample, possibly resulting falsely negative in subjects undergoing concomitant antibiotic treatment or a false positive result can be found by contamination. The methods based on molecular biology do not require living germs and, therefore, are not characterised by the sensitivity limitations that are typical of cultural methods. For this reason, such methods can result to be extremely effective in patients who have already received an antibiotic therapy, and are not affected by rapid transport (so much so that samples can be stored at room temperature even for a few days) and, finally, do not require any culture medium.

In the present study, when an infant has to undergone blood sample for bacteria culture to verify a possible sepsis, a residual blood (200µl) is processed in the same time using a kit based on molecular biology. This kit is designed to obtain the highest sensitivity and specificity in the determination of most invasive bacterial diseases (meningitis, sepsis, pneumonia, etc.) affecting full-term, preterm infants to determine any presence of bacterial DNA belonging to all serotypes of Klebsiella pneumoniae, Escherichia coli, Streptococcus agalactiae and Listeria monocytogenes The target bacteria have been chosen on the basis of the current Italian epidemiological context, so as to include germs causing about 90% of the meningitis/sepsis cases among the neonatal population. The detection system can unmistakably identify the germ against which it is directed and without causing any cross-reaction with other germs or human DNA.

The results obtained with this method have demonstrated a 100% specificity (no false positive result). The sensitivity of this method compared with the cultural method has turned out to be twice as high.

The aim of the present study is to compare the efficacy of the blood culture method and the kit for molecular detection of bacterial DNA (all serotypes of Klebsiella pneumoniae, Escherichia coli, Streptococcus agalactiae and Listeria monocytogenes) considering the relevant epidemiology of our NICU, in order to verify the relative frequency of neonatal sepsis (EOS and LOS) caused by the target bacteria on the whole frequency of the bacteria responsible of all the sepsis in our ward.

The observational estimated period to collect 100 measurable samples, is 18 months from the beginning of the enrolment.

Samples correspond to the enrollment of term o preterm neonates who needed a blood withdrawal for a suspect of sepsis, that are processed by both mothods.

ELIGIBILITY:
Infants with: suspected Blood stream infection, hospitalized in the NICU, with SIRS ≥2.

Exclusion Criteria: infants with genetic and/or congenital diseases, parents refusing to sign a written informed consent.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (full-term or pre-term) requiring to be sampled for suspected sepsis (EOS or LOS)
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
frequency of positive test | 1 week
  to verify the frequency of positive test (neonatal sepsis, EOS or LOS) detected by the molecular assay compare to these of the blood culture

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Stronati, MD, Study Director — Fondazione IRCCS Policlinico S. Matteo, 27100 Pavia Italy
Locations (1):
- Neonatal Unit, IRCCS Policlinico S. Matteo., Pavia, PV, Italy

REFERENCES:
- [Background] • Istituto Superiore di Sanità. http//www.simi.iss.it/dati.htm • Shah BA, Neonatal sepsis: an old problem with new insights PadburyJF. Virulence 5:1, 163-171; January 1, 2014; © 2014 • Stoll BJ, Hansen NI, Sánchez PJ, Faix RG, Poindexter BB, Van Meurs KP, Bizzarro MJ, Goldberg RN, Frantz ID 3rd, Hale EC, et al.; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Early onset neonatal sepsis: the burden of group B Streptococcal and E. coli disease continues. Pediatrics 2011; 127:817-26. • Libster R, Edwards KM, Levent F, Edwards MS, Rench MA, Castagnini LA, Cooper T, Sparks RC, Baker CJ, Shah PE. Long-term outcomes of group B streptococcal meningitis. Pediatrics 2012; • Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, et al. Late-onset sepsis in very low birth weight neonates: the experience of the NICHD Neonatal Research Network. Pediatrics 2002; 110:285-91; • Levy MM, Fink MP, Marshall JC et al. "2001 SCCM/ESICM/ACCP ATS/SIS International Sepsis Definitions Conference" Critical Care Medicine . 31 n 4 pp: 1250-1256, 2003. • Arnon S. Litmanovitz I. Diagnostic tests in neonatal sepsis. Curr Opinion Infectious Dis 2008; 21: 223-27. • Russell JA. Management of sepsis. N Engl J Med 2006;355:1699-713. • Overturf GD. Defining bacterial meningitis and other infections of the central nervous system. Pediatr Crit Care Med. 2005;6(3 Suppl):S14-8.
- [Derived] Mazzucchelli I, Garofoli F, Angelini M, Tinelli C, Tzialla C, Decembrino L. Rapid detection of bacteria in bloodstream infections using a molecular method: a pilot study with a neonatal diagnostic kit. Mol Biol Rep. 2020 Jan;47(1):363-368. doi: 10.1007/s11033-019-05138-2. Epub 2019 Oct 22. PMID 31642041